CLINICAL TRIAL: NCT05194059
Title: ActiPacMAN: 'Activity Pacing' in PLWH With Fatigue Symptoms. Monitoring Through the Combined Use of Actigraphy and Mobile App Notifications
Brief Title: 'Activity Pacing' in PLWH With Fatigue Symptoms.
Acronym: ActiPacMAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Scientific Institute San Raffaele (Other)
Responsible Party: Principal Investigator, Paola Cinque, Principal Investigator, Scientific Institute San Raffaele
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ActiPacMAN
Record Dates: First submitted 2022-01-03; First posted 2022-01-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Hiv
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Participants will follow a personalized activity pacing program for 16 weeks with the support of a heath band and a mobile application for tablet
  Interventions: Behavioral: Home-based physical activity
- Control Group (No Intervention): Participants will follow a personalized activity pacing program for 16 weeks without any other support

INTERVENTIONS:
Behavioral: Home-based physical activity — Participants will follow a personalized activity pacing program
  Arms: Experimental Group

SUMMARY:
Physical activity helps to improve health and prevent chronic diseases. However, the fatigue usually hampers the training and execution of physical exercises, especially in people with chronic fatigue syndromes (CFCs), such as persons living with HIV (PLWH). We hypothesize that the "activity pacing", i.e. the strategy to optimize daily physical activity into manageable exercises in a way that should not exacerbate fatigue symptoms, may help a progressive improvement in physical activity of a group of PLWH with fatigue symptoms. Motivation and adherence to exercise will be monitored through the use of digital supports.

ELIGIBILITY:
Inclusion Criteria:

* of age ≥18 years;
* either sedentary or already practicing mild/moderate physical activity (at least 150 minutes of moderate-intensity physical activity throughout the week);
* able to sign the informed consent.

Exclusion Criteria:

The study will exclude HIV+ individuals:

* with any HIV-related disease requiring hospitalization in the 6 weeks before enrolment;
* with medical conditions (e.g. neurologic, muscular-skeletal, cardiovascular diseases) contraindicating non agonistic exercise, as established by a sport medicine specialist;
* currently abusing of substance or alcohol;
* already performing physical activity at higher level than the current WHO recommendations (30 minutes of moderate activity 5 times a week).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-12-03 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2022-10-28 (Actual)

PRIMARY OUTCOMES:
Activity pacing improvement | 16 week
  To compare the improvement in the physical fitness between the Experimental Group and Control Group

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Infectious Diseases, Milan, Italy

IPD SHARING:
Plan to Share IPD: Yes